CLINICAL TRIAL: NCT01410448
Title: A 3-month, Multicenter, Randomized, Open Label Study to Evaluate the Impact of Early Versus Delayed Introduction of Everolimus on Wound Healing in de Novo Kidney Transplant Recipients With a Follow-up Evaluation at 12 Month After Transplant (NEVERWOUND Study)
Brief Title: Everolimus in de Novo Kidney Transplant Recipients
Acronym: NEVERWOUND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AIT25; 2011-002866-19 (EudraCT Number)
Record Dates: First submitted 2011-08-02; First posted 2011-08-05 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplantation
Keywords: Immunosuppression; Kidney transplantation; everolimus; safety
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Cyclosporine; Steroids

ARMS (2):
- Immediate Everolimus (IE) (Active Comparator): Everolimus was started within 48 hours after graft reperfusion at a starting dose of 0.75 mg twice daily in combination with low-dose cyclosporine and steroids for 3 months.
  Interventions: Drug: Everolimus; Drug: Cyclosporine; Drug: Steroids
- Delayed Everolimus (Experimental): The standard dose of mycophenolate sodium was administered within 48 hours after graft reperfusion in combination with a full dose of cyclosporine and steroids. After28 +/- 4 days of treatment, mycophenolate sodium was discontinued and everolimus was introduced at a starting dose of 0.75 mg twice daily for 3 months.
  Interventions: Drug: Everolimus; Drug: Mycophenolate sodium; Drug: Cyclosporine; Drug: Steroids

INTERVENTIONS:
Drug: Everolimus — Everolimus was provided in blisters containing 0.25 and 0.75 mg tablets and was taken orally.
  Other Names: Certican®
Drug: Mycophenolate sodium — Two 360 mg tablets were administered twice daily at 12-hour intervals. The tablets were swallowed whole in order to maintain the integrity of the enteric coating.
  Other Names: Myfortic®
  Arms: Delayed Everolimus
Drug: Cyclosporine — Cyclosporine was supplied as blisters containing 100 mg, 50 mg, 25 mg and 10 mg soft-gelatin capsules and was administered orally.
  Other Names: Neoral®
Drug: Steroids — Steroids were administered according to local clinical practice.

SUMMARY:
The purpose of this study was to evaluate whether delayed (i.e. 28 ± 4 days post-transplant) administration of everolimus after transplantation reduces the risk of wound healing complications in comparison with immediate administration in de novo renal transplant patients (proportion of patients without wound/surgical complications related to initial transplant surgery) between randomization and 3 months after transplantation.

ELIGIBILITY:
Key Inclusion criteria:

* Patients who are willing and able to participate in the study and who provide written informed consent before performing any study related procedure;
* Men or women ≥18 years at transplant;
* Recipients of 1st or 2nd single kidney transplant from deceased donor or living unrelated/related donor > 14 years;

Key Exclusion criteria:

* Patients who are recipients of multiple organs transplant, including two kidneys;
* Historical or current peak PRA > 50%. Patients with already existing antibodies against the donor;
* Thrombocytopenia (platelets < 75,000/mm³), absolute neutrophil count <1,500/mm³, leucopenia (leucocytes < 2,500/mm³) or hemoglobin < 7 g/dL;
* Body mass index (BMI) > 30 Kg/m2;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- Italy (18):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Coppito, AQ
  - Novartis Investigative Site, Bari, BA
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Siena, SI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Novara

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included a 3 month treatment period followed by an observational follow-up period. Participants were treated as per local practice during follow-up and a follow-up evaluation was performed at 12 months.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to one of the 2 treatment groups.
Groups:
- Delayed Everolimus (DE): The standard dose of mycophenolate sodium was administered within 48 hours after graft reperfusion in combination with a full dose of cyclosporine and steroids. After28 +/- 4 days of treatment, mycophenolate sodium was discontinued and everolimus was introduced at a starting dose of 0.75 mg twice daily for 3 months.
Period: Overall Study
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Started | 193 | 190
Intent-to Treat (ITT) Analysis Set | 193 | 190
Modified ITT Analysis Set | 161 | 149
Completed | 181 | 155
Not Completed | 12 | 35
Not completed — No conversion to everolimus | 0 | 24
Not completed — Graft loss | 4 | 1
Not completed — Administrative issues | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Protocol Violation | 0 | 4
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE) | Total
Number analyzed (Participants) | 193 | 190 | 383
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.46 (11.37) | 51.19 (12.29) | 51.32 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 58 | 117
  Male | 134 | 132 | 266

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Wound Healing Complications - Worst-case Scenario
Description: The percentage of participants without wound healing complications was assessed. Wound healing complications consisted of lymphorrhea, fluid collections, wound dehiscence, wound infections and incisional hernia. In the worst-case scenario, failure, i.e. at least one healing complication occurrence, was identified in one of the following cases: wound complication occurrence, missing information about wound complication occurrence, or study discontinuation due to any reason.
Time Frame: 3 months
Population: The safety population, which included all randomized participants who were treated and had at least one safety assessment, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 68.39 | 61.58
Statistical Analysis 1: Comparison: Immediate Everolimus (IE) vs Delayed Everolimus (DE); Test type: Superiority or Other; p = 0.0921, Regression, Logistic

2. Secondary Outcome: Percentage of Participants Without Wound Healing Complications - Worst-case Scenario
Description: The percentage of participants without wound healing complications was assessed. Wound healing complications consisted of lymphorrhea, fluid collections, wound dehiscence, wound infections and incisional hernia. In the worst-case scenario, failure, i.e. at least one healing complication occurrence, was identified in one of the following cases: wound complication occurrence, missing information about wound complication occurrence or study discontinuation due to any reason for participants who did not complete the 12 month follow-up visit.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 65.80 | 59.47

3. Secondary Outcome: Percentage of Participants Who Experienced Treatment Failure - Worst-case Scenario
Description: The percentage of participants who experienced treatment failure was assessed. Treatment failure was defined as the occurrence of at least one failure event among death, graft loss or biopsy-proven acute rejection (BPAR). In the worst-case scenario, treatment failure was identified in one of the following cases: occurrence of at least one treatment failure event or study discontinuation due to any reason.
Time Frame: 3 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 11.40 | 21.05

4. Secondary Outcome: Patient Survival Rate: Percentage of Deaths - Worst-case Scenario
Description: The percentage of deaths was assessed. In the worst-case scenario, failure, i.e. death, was identified in one of the following cases: participant's death or study discontinuation due to any reason.
Time Frame: 3 Months, 12 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 6.22 | 18.42

5. Secondary Outcome: Participant/Graft Survival Rate: Percentage of Participants With Failure Events of Death or Graft Loss - Worst-case Scenario
Description: The percentage of participants who experienced death or graft loss was assessed. In the worst-case scenario, failure, i.e. participants death or graft loss, was identified in one of the following cases: occurrence of at least one failure event or study discontinuation due to any reason.
Time Frame: 3 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 6.74 | 18.42

6. Secondary Outcome: Graft Survival Rate: Percentage of Participants With Graft Loss - Worst-case Scenario
Description: The percentage of participants who experienced graft loss was assessed. In the worst-case scenario, failure, i.e. graft loss, was identified in one of the following cases: occurrence of graft loss or discontinuation due to any reason.
Time Frame: 3 months, 12 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants
  3 months | 6.74 | 18.42
  12 months | 7.25 | 19.47

7. Secondary Outcome: Percentage of Participants With BPAR - Worst-case Scenario
Description: A biopsy-proven acute rejection was defined as a biopsy graded IA, IB, IIA, IIB or III. In the worst-case scenario, failure, i.e. BPAR, was identified in one of the following cases: occurrence of BPAR or study discontinuation due to any reason.
Time Frame: 3 Months, 12 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants
  3 monts | 11.40 | 21.05
  12 months | 15.54 | 24.74

8. Secondary Outcome: Percentage of Participants With Delayed Graft Function (DGF) -
Description: DGF was defined as the need for dialysis in the first week after transplant, excluding Renal Replacement Therapy within the first 24 hours after transplantation.
Time Frame: 3 Months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 23.83 | 31.58

9. Secondary Outcome: Duration of DGF
Description: The duration of DGF was defined as the elapsed time from first to last day of post-transplant dialysis.
Time Frame: 3 months
Population: Participants from the Intent-to-Treat (ITT) populations who required dialysis, 46 (23.83%) of the IE group and 60 (31.58%) of the DE group, were analyzed. The ITT population included all randomized participants who were treated.
Measure: Median (Full Range); unit: Days
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 46 | 60
Days | 8.50 [1 to 93] | 5.50 [1 to 76]

10. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) (Calculated With Modified Diet in Renal Disease (MDRD)-4 Formula - ITT
Description: Renal function was assessed by measuring serum creatinine and serum urea and by calculating creatinine clearance using the MDRD-4 formula. eGFR = 186.3*(serum creatinine [mg/dL])^-1.154 * (age at screening) -0.203 * (0.742 if female) * (1.21 if African American). A positive change from baseline indicates improvement.
Time Frame: baseline, 3 Months
Population: Participants from the ITT, who had both baseline and month 3 measurements, were included in the analysis for the month 3 time point. The ITT population included all randomized participants who were treated.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 187 | 183
mL/min | 38.64 (22.45) | 39.13 (21.46)

11. Secondary Outcome: Change From Baseline in Estimated Glomerular Filtration Rate (eGFR) (Calculated With Modified Diet in Renal Disease (MDRD)-4 Formula - Modified ITT
Description: as for outcome 10
Time Frame: baseline, 12 months
Population: Participants from the modified ITT, who had both baseline and month 12 measurements, were included in the analysis for the month 12 time point. The modified ITT included participants who completed the Core Phase (at 3 months) without discontinuing the treatment and performed the subsequent follow-up evaluation at 12 months after transplant.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 151 | 142
mL/min | 41.26 (18.69) | 41.56 (19.90)

12. Secondary Outcome: Change From Baseline in Serum Creatinine - ITT
Description: Blood samples were collected to assess serum creatinine measurements. A negative change from baseline indicates improvement.
Time Frame: baseline, 3 months
Population: Participants from the ITT, who had both baseline and the post-baseline measurement for a given post-baseline time point, were included in the analysis for that post-baseline time point. The ITT population included all randomized participants who were treated.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 187 | 183
mg/dL | -4.79 (2.74) | -5.13 (2.32)

13. Secondary Outcome: Change From Baseline in Serum Creatinine - Modified ITT
Description: as for outcome 12
Time Frame: baseline, 12 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 150 | 141
mg/dL | -4.96 (2.48) | -5.22 (2.24)

14. Secondary Outcome: Percentage of Participants With Proteinuria
Description: Incidence of proteinuria (>1,000 mg/day in urine collected in 24 hours or > 1.0 if measured on the urine protein/creatinine concentration ratio in a spot urine sample) was assessed.
Time Frame: 3 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants
  Yes | 4.15 | 4.21
  No | 68.91 | 68.42
  Missing | 26.94 | 27.37

15. Secondary Outcome: Percentage of Participants With Acute Rejection (AR)
Description: AR was defined as an episode of increased serum creatinine >30% that was clinically diagnosed as an acute rejection but was not biopsy proven.
Time Frame: 12 months
Population: The intent to treat (ITT) population, which included all randomized participants who were treated, was analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 193 | 190
Percentage of participants | 12.44 | 10.53

16. Secondary Outcome: Percentage of Participants With a New Onset of Malignancy
Description: The percentage of participants with a new onset of malignancy was assessed.
Time Frame: 12 months
Population: Participants from the modified ITT, who had values at 12 months, were analyzed. The modified ITT included participants who completed the Core Phase (at 3 months) without discontinuing the treatment and performed the subsequent follow-up evaluation at 12 months after transplant.
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 159 | 147
Percentage of participants | 0 | 0.68

17. Secondary Outcome: Percentage of Participants With a New Onset of Diabetes
Description: The percentage of participants with a new onset of diabetes was assessed.
Time Frame: 12 months
Population: as for outcome 16
Measure: Number; unit: Percentage of participants
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Number analyzed (Participants) | 159 | 148
Percentage of participants | 3.14 | 4.05

ADVERSE EVENTS:
Arm/Group | Immediate Everolimus (IE) | Delayed Everolimus (DE)
Serious Adverse Events (participants affected / at risk) | 73/193 | 61/190
Other Adverse Events (participants affected / at risk) | 155/193 | 156/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Everolimus (IE) (N=193) | Delayed Everolimus (DE) (N=190)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Protein S deficiency (Congenital, familial and genetic disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 2 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 2 | 0
Hyperpyrexia (General disorders) | 1 | 1
Impaired healing (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 11 | 4
Transplant rejection (Immune system disorders) | 3 | 1
Abscess (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 3
Device related infection (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Renal abscess (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 8 | 7
Urosepsis (Infections and infestations) | 1 | 2
Wound infection (Infections and infestations) | 3 | 2
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 | 3
Expired product administered (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Graft loss (Injury, poisoning and procedural complications) | 3 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 0 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 1
Perinephric collection (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Renal transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Ureteric anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 2
Blood creatinine increased (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 2 | 0
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Perinephric effusion (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 2
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal artery thrombosis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Renal impairment (Renal and urinary disorders) | 3 | 2
Renal ischaemia (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Renal vein thrombosis (Renal and urinary disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Urinary fistula (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinoma (Renal and urinary disorders) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bladder catheter replacement (Surgical and medical procedures) | 1 | 0
Lymphocele marsupialisation (Surgical and medical procedures) | 1 | 1
Arterial thrombosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 7 | 7
Lymphorrhoea (Vascular disorders) | 0 | 2
Shock (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Immediate Everolimus (IE) (N=193) | Delayed Everolimus (DE) (N=190)
Anaemia (Blood and lymphatic system disorders) | 67 | 58
Leukopenia (Blood and lymphatic system disorders) | 8 | 14
Abdominal pain (Gastrointestinal disorders) | 14 | 15
Constipation (Gastrointestinal disorders) | 12 | 13
Nausea (Gastrointestinal disorders) | 4 | 14
Oedema peripheral (General disorders) | 17 | 14
Pyrexia (General disorders) | 16 | 14
Cytomegalovirus infection (Infections and infestations) | 13 | 16
Urinary tract infection (Infections and infestations) | 34 | 34
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 26 | 23
Dyslipidaemia (Metabolism and nutrition disorders) | 28 | 24
Hypercholesterolaemia (Metabolism and nutrition disorders) | 20 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 10 | 18
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 10
Hyperphosphataemia (Metabolism and nutrition disorders) | 20 | 13
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 14 | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 21 | 25
Hypocalcaemia (Metabolism and nutrition disorders) | 24 | 30
Hypokalaemia (Metabolism and nutrition disorders) | 26 | 24
Haematuria (Renal and urinary disorders) | 14 | 3
Haematoma (Vascular disorders) | 12 | 6
Hypertension (Vascular disorders) | 34 | 30
Lymphocele (Vascular disorders) | 25 | 33
Lymphorrhoea (Vascular disorders) | 6 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.